CLINICAL TRIAL: NCT00202332
Title: A Prospective Randomised Study od Coronary Artery Bypass Surgery Without the Use of Cardiopulmonary Bypass
Brief Title: CABG Without the Use of CPB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1999.115
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Bypass
MeSH Terms: interventions — Coronary Artery Bypass

INTERVENTIONS:
Procedure: Coronary artery bypass

SUMMARY:
Comparison of clinical outcomes in patients undergoing coronary bypass surgery using the heart/lung machine as opposed to using off-pump techniques.

ELIGIBILITY:
Inclusion Criteria: Eligible for coronary surgery -

Exclusion Criteria: Less than 18 years Emergency and salvage operations

-

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2003-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Comparison of clinical outcomes for coronary artery bypass graft surgery when performed using cardiopulmonary bypass versus beating heart surgery without cardiopulmonary bypass | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Davis, MD, Study Chair — Melbourne Health